CLINICAL TRIAL: NCT01216124
Title: A Prospective, Open and Unicentric Phase II Clinical Trial of Docetaxel Combined With Oxaliplatin for Triple Negative Local Advanced Breast Cancer Patients (TNLABC)
Brief Title: Efficacy and Safety Study of Neoadjuvant Chemotherapy for Local Advanced Triple Negative Breast Cancer Patients
Status: Available | Type: Expanded Access
Sponsor: Fudan University (Other)
Collaborators: Chinese Anti-Cancer Association (Other)
Responsible Party: Chinese Anti-Cancer Association，Committee Breast Cancer Society
Other Study IDs: Fudan TNBC Neo CT
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2009-09

CONDITIONS: Triple Negative Local Advanced Breast Cancer
Keywords: triple negative local advanced breast cancer(TNLABC),neoadjuvant chemotherapy

INTERVENTIONS:
Drug: docetaxel oxaliplatin — docetaxel 75mg/m2 D1 oxaliplatin 130mg/m2 D2
  1 cycle=21 days DO*6

SUMMARY:
The 10%-15% of breast carcinomas known to be 'triple negative (TN)' (not expressing HRs and not exhibiting overexpression Her2) constitutes 85% of all basal-like tumors, because it is based on three standard immunohistochemical biomarkers.

In clinical routine, Docetaxel was widely indicated as first-line therapy for breast cancer patients in adjuvant or neoadjuvant settings. Oxaliplatin, trans-1-diaminocyclohexane-platinum, may offer advantages over other platinum agents. Oxaliplatin promotes formation of DNA adducts, preventing DNA replication and transcription and ultimately causing apoptosis. Oxaliplatin was more potent than cisplatin and the Oxaliplatin-based regimen was active for the patients of lung cancer, colorectal cancer and ect. TNBC patients were more sensitive to platinum-based chemotherapy regimens according to the results of some retrospective studies. There was no report about Oxaliplatin in the chemotherapy setting for breast cancer patients.

The investigators hypothesized that using Oxaliplatin adding to docetaxel would be feasible and active in patients with TNLABC because in vitro findings suggest synergism between the agents. This study was designed to investigate the efficacy and toxicity of oxaliplatin-based regimen as a neoadjuvant chemotherapy setting in triple negative local advanced breast cancer patients

DETAILED DESCRIPTION:
Eligibilty Female adults(>18 years old) were eligible if they had histologically or cytologically confirmed stage IIIb or IIIc TNLABC that had not been treated with any systemic treatment. Patients also had Eastern Cooperative Oncology Group(ECOG) Performance status of 0 or 1, absolute neutrophil count (ANC)>1500/mm3,hemoglobin >8.0g/dL, and platelet count >100,000/mm3,creatinine<2.5 times the upper limit of normal(ULN)）, transaminases<2.5 times ULN or alkaline phosphatase<4 times ULN if transaminases was normal, and total bilirubin <2.5 times ULN. Exclusion criteria were active infection, pregnancy, other primary malignancy (except in situ carcinoma of cervix or adequately treated nonmelanomatous carcinoma of the skin), any documented distant metastasis and uncontrolled systemic diseases.

This study protocol was approved by institutional ethic review boards and conducted according to guidelines for good clinical practice and the Helsinki Declaration.All patients provided written informed consent.

Study design and treatment plan This was a prospective, open and unicentric phase II clinical study. All chemotherpy was administered intravenously on an outpatient basis. The patients received dexamethasone 7.5mg orally twice a day for 3 days before the day of chemotherapy. On day 1, docetaxel 75mg/m2 was infused over 60 minutes as well as oxaliplatin 130mg/m2 was infused over 120 minutes on day 2. Thirty minutes before chemotherapy, premedication consisted of a 5-hydroxytryptamine3(HT3) receptor antagonist. Furthermore, Vitamin C 2g and Vitamin B2 200mg were followed immediately after the chemotherapy. Treatment was administered every 21 days for a maximum of four cycles or until disease progression or unacceptable toxicity.The prophylactic use of a colony-stimulating factor (CFS) was not permitted in the first cycle.

An initial diagnosis of unilateral primary breast cancer without distant metastases, at least 7 months of follow-up information for disease recurrence and death and triple receptor negative for estrogen receptor (ER), progesterone receptor (PR), Her2 were included as pre-treatment evaluation. Moreover tumor size, number of involved axillary lymph nodes (ALN), clinical stage and biomarkers such as Cathepsin-D, P53, nm23, PS2 and PCNA, were recorded as available information for further analysis. In the procedure of neoadjuvant chemotherapy, weekly or biweekly complete blood cell counts, physical examination, electrocardiogram (EKG), liver and rental function tests should be repeated. Tumor size was assessed by magnetic resonance imaging (MRI) every two cycles or when the clinical signs suggested disease progression as well as before the chemotherapy. Tumor response was determined by response evaluation criteria in solid tumors (RECIST). Complete and partial response (CR and PR) should be confirmed on two assessments performed at least four weeks apart.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged from 18 to 65 years;
2. Histologically or cytologically proven invasive unilateral breast cancer (regardless of the type);
3. Initial clinical condition compatible with complete initial resection;
4. No residual macro or microscopic tumor after surgical excision;
5. Patient presenting one of the following criteria (reviewed before randomization by referent pathologist):

   Triple Negative(ER-PR-Her-2-) Hormone receptor negativity is defined as ER<10%, PR<10% (IHC), HER2 negativity is defined as IHC 0-1+, or [IHC 2+ and FISH or CISH negative].
6. No clinically or radiologically detectable metastases (M0);
7. No peripheral neuropathy > 1;
8. WHO Performance status (ECOG) of 0 or 1;
9. Adequate hematological function (neutrophil count ³ 2x109/l, platelet count ³ 100x 109/l, Hemoglobin > 9 g/dl);
10. Adequate hepatic function: ASAT and ALAT £ 1.5 ULN alkaline phosphatases £ 2.5 ULN,total bilirubin £ 1,5 ULN;
11. Adequate renal function: serum creatinine £ 1.5 ULN;
12. Patients accepting contraception intake during the overall length of treatment if of childbearing potential;
13. Adequate cardiac function, LEVF value > 50% by Muga scan or echocardiography;
14. Signed written informed consent.

Exclusion Criteria:

1. Bilateral breast cancer or patient with controlateral DCIS;
2. Any metastatic impairment, including homolateral sub-clavicular node involvement,regardless of its type;
3. Any tumor ³ T4a (UICC1987) (cutaneous invasion, deep adherence, inflammatory breast cancer);
4. Luminal A, Luminal B and Her-2 overexpression
5. Any clinically or radiologically suspect and non-explored damage to the controlateral breast;
6. Previous cancer (excepted cutaneous baso-cellular epithelioma or uterine peripheral epithelioma) in the preceding 5 years, including invasive controlateral breast cancer;
7. Patients already included in another therapeutic trial involving an experimental drug;
8. Patients with other concurrent severe and/or uncontrolled medical disease or infection which could compromise participation in the study;
9. LEVF < 50% (MUGA scan or echocardiography);
10. Clinically significant cardiovascular disease (e.g. unstable angina, congestive heart failure, uncontrolled hypertension (>150/90), myocardial infarction or cerebral vascular accidents) within 6 months prior to randomization;
11. Known prior severe hypersensitivity reactions to agents in this study
12. Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and up to 8 weeks after treatment completion;

14) Women who are pregnant or breastfeeding. Adequate birth control measures should be taken during study treatment phase; 15) Women with a positive pregnancy test en enrollment or prior to study drug administration; 16) Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial; 17) Individual deprived of liberty or placed under the authority of a tutor.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult